CLINICAL TRIAL: NCT01734876
Title: Short and Long-term Effects of Tactile Touch on Salivary Cortisol Concentrations in Parkinson's Disease.
Brief Title: Effects of Tactile Touch on Chronic Pain in Parkinson´s Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Jönköping County (Other Government)
Collaborators: University Hospital, Linkoeping (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D 03-673; FUTURUM 254481 (Other Grant/Funding Number: FUTURUM 254481)
Record Dates: First submitted 2012-11-11; First posted 2012-11-28 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2012-11

CONDITIONS: Pain; Sleep
Keywords: Parkinson´s disease; Pain; Sleep; HPA axis function; Health Related Quality of Life
MeSH Terms: conditions — Pain; Parkinson Disease | interventions — Touch; Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tactile Touch (Experimental): Tactile Touch is given to the active arm
  Interventions: Behavioral: Tactile Touch; Behavioral: Rest To Music
- Rest To Music (Active Comparator): Rest to Music. Rest for 30-60 minutes, aroma therapy, quit music in the background, well temepered room, lying position
  Interventions: Behavioral: Tactile Touch; Behavioral: Rest To Music

INTERVENTIONS:
Behavioral: Tactile Touch — Tactile Touch was performed for 10 times during a 8 week period.The method consists of a superficial whole body tactile touch, following a structural scheme. Participants in a horizontal position, in a tempered room. Aroma of lavendar and quiet music in the background.
  Other Names: massage therapy
Behavioral: Rest To Music — Participants in horizontal position. Rest in a temperated room, aromas and quiet music in the background. Time: About 30 minutes.

SUMMARY:
The Parkitouch study compared the effects on pain, sleep quality and HealthRelated Quality of Life (HRQoL) among 44 participants with Parkinson´s Disease for at least two years and chronic pain.The two groups were randomized to either Tactile Touch and Rest to Music or only Rest to Music alone. It was prospective and had a duration of 34 weeks. The first 10 weeks was the intervention period , followed by a follow-up period. Outcome measures were salivary cortisol concentration measured at seven occasions of which two were immediately before, after and 30 minutes after intervention. Diurnal salivary cortisol was calculated based on four timepoints of sampling per 24 hour period.

DETAILED DESCRIPTION:
This study was initiated by the massage therapists who had experienced pain reduction in parkinsonian patients when usin Tactile Touch. As the method consisted of a combination of Music Therapy and Aroma therapy we chose just to study the effects of the Tactile Touch.

HrQOL was measured using SF-36 (Swe.ver.1) sleep was measured with the PDSS scale, pain wit VAS 10 cm scale and the Pain-O.Meter. All measures were repeated during the study period.

Patients were not allowed to change their basic antiparkinson medication.All drugs were carefully registered and supervised by specialists in neurology at the three different study sites in Southern Sweden. The massage technique was described in a 11 A4 pages long description and the same method was used at all three sites. The same aroma oils, same temperature in the rooms and the same music was used.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson´s Disease
* chronic pain

Exclusion Criteria:

* Epilepsy
* Active malignancy
* Diabetes mellitus
* Parkinson´s disease in complication phase

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-09; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Effect of Tactile Touch on Hypothalamo Pituitary Adrenal (HPA) axis function in Parkinson Disease with chronic pain | Within 1 year
  HPA axis function in PD patients (salivary cortisol, mmol / l diurnal curve , pre and post intervention).

SECONDARY OUTCOMES:
Effect of Tactile Touch on HRQoL | Within 1 year
  As secondary endpoints, HealthRelated Quality of Life (HRQoL),measured by SF-36,Swe ver.1 sleep quality measured by Parkinson Disease Sleep Scale (PDSS)

OTHER OUTCOMES:
The Parkitouch Study | Wihin 1 year
  Are Tactile Touch more effective than Rest to Music in reducing patients´ chronic stress in terms of lowering salivary cortisol secretion in short and / or long term perspective? Is the treatment safe and well tolerated? Does sleep quality improve and is sleep fragmentaion reduced? Is HRQoL improved?

CONTACTS AND LOCATIONS:
Overall Officials: Carl Jo Törnhage, MD, PhD, Principal Investigator
Locations (1):
- FUTURUM, Jönköping, Sweden

REFERENCES:
- [Result] Skogar O, Fall PA, Hallgren G, Lokk J, Bringer B, Carlsson M, Lennartsson U, Sandbjork H, Tornhage CJ. Diurnal salivary cortisol concentrations in Parkinson's disease: increased total secretion and morning cortisol concentrations. Int J Gen Med. 2011;4:561-9. doi: 10.2147/IJGM.S20875. Epub 2011 Aug 10. PMID 21887109
- [Result] Skogar O, Fall PA, Hallgren G, Bringer B, Carlsson M, Lennartsson U, Sandbjork H, Tornhage CJ, Lokk J. Parkinson's disease patients' subjective descriptions of characteristics of chronic pain, sleeping patterns and health-related quality of life. Neuropsychiatr Dis Treat. 2012;8:435-42. doi: 10.2147/NDT.S34882. Epub 2012 Oct 12. PMID 23091387
- [Derived] Tornhage CJ, Skogar O, Borg A, Larsson B, Robertsson L, Andersson L, Andersson L, Backstrom P, Fall PA, Hallgren G, Bringer B, Carlsson M, Lennartsson UB, Sandbjork H, Lokk J. Short- and long-term effects of tactile massage on salivary cortisol concentrations in Parkinson's disease: a randomised controlled pilot study. BMC Complement Altern Med. 2013 Dec 13;13:357. doi: 10.1186/1472-6882-13-357. PMID 24330473
- See also: Parkinson's disease patients' subjective descriptions of characteristics of chronic pain, sleeping patterns and Health Related Quality of Life — http://www.ncbi.nlm.nih.gov/pubmed?term=Parkinson%E2%80%99s%20disease%20patients%E2%80%99%20subjective%20descriptions%20of%20characteristics%20of%20chronic%20pain%2C%20sleeping%20patterns%20and%20Health%20Related%20Quality%20of%20Life
- See also: Diurnal salivary cortisol concentrations in Parkinson's disease: increased total secretion and morning cortisol concentrations — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3160865/